CLINICAL TRIAL: NCT06678646
Title: Ultrasound-guided Release of the Median Nerve at the Elbow in Patients With Lacertus Syndrome
Acronym: LACECHOCHIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A01191-46
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Median Nerve Entrapment
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound guided surgery (Experimental): Percutaneous Ultrasound-Guided Release of the Lacertus Fibrosus for Median Nerve Entrapment at the Elbow
  Interventions: Procedure: Elbow ultrasound-guided surgery

INTERVENTIONS:
Procedure: Elbow ultrasound-guided surgery — Percutaneous Ultrasound-Guided Release of the Lacertus Fibrosus for Median Nerve Entrapment at the Elbow

SUMMARY:
Lacertus syndrome is an orthopaedic condition that occurs when the median nerve is compressed where it passes under the lacertus fibrosus.

Treatment for lacertus syndrome is generally aimed at relieving compression of the median nerve and reducing associated symptoms. Treatment options vary according to the severity of the condition and the patient's individual needs.

Sectioning the Lacertus fibrosus frees the median nerve. It is performed as an outpatient procedure under local anaesthetic, and the patient can resume his or her activities immediately. Lacertus fibrosus section has been described as an open procedure, i.e. with a horizontal scar in the elbow crease.

Ultrasound guided surgery is an innovative technique that has proved its effectiveness for nerve releases such as the median nerve in the carpal tunnel or the ulnar nerve in the elbow. This technique was tested on a series of 18 cadavers and then on a series of 15 patients with a lacertus syndrome. The patients underwent the operation without any immediate surgical or anaesthetic complications. Muscle strength returned immediately and persisted. Pain was reduced and all patients who were working were able to carry out their professional activities from the very first week. The millimetric skin incision healed without hypertrophic scar tissue. A small haematoma appeared at week 1 and resolved spontaneously. No other late complications were observed.

In this context, this study would consolidate the preliminary results observed and confirm the hypothesis that minimally invasive percutaneous surgery under ultrasound is appropriate for sectioning Lacertus fibrosus safely, rapidly and effectively in Lacertus syndrome.

DETAILED DESCRIPTION:
The lacertus fibrosus is a thick, tough, fibrous band of connective tissue. The lacertus fibrosus is a continuation of the tendon of the biceps brachii muscle. It plays a role in protecting the median nerve, which passes under this ligament as it travels towards the hand.

Lacertus syndrome is an orthopaedic condition that occurs when the median nerve is compressed where it passes under the lacertus fibrosus. This syndrome can affect both men and women, generally after the age of 35. It can occur on one side or bilaterally. Common symptoms vary from person to person and include pain in the forearm, elbow and sometimes the shoulder, a feeling of tiredness or heaviness in the forearm, muscle weakness in the thumb and grip, clumsiness, loss of stamina and variable tingling in the first three fingers of the hand (thumb, index and middle fingers), similar to carpal tunnel syndrome.

Treatment for lacertus syndrome is generally aimed at relieving compression of the median nerve and reducing associated symptoms. Treatment options vary according to the severity of the condition and the patient's individual needs. They may include physiotherapy, non-steroidal anti-inflammatory drugs (NSAIDs), orthoses, corticosteroid injections and surgery.

Sectioning the Lacertus fibrosus frees the median nerve. It is performed as an outpatient procedure under local anaesthetic, and the patient can resume his or her activities immediately. Lacertus fibrosus section has been described as an open procedure, i.e. with a horizontal scar in the elbow crease.

Ultrasound guided surgery is an innovative technique that has proved its effectiveness for nerve releases such as the median nerve in the carpal tunnel or the ulnar nerve in the elbow. This new ultrasound-guided surgical technique reduces the side-effects associated with surgery (infection, algodystrophy, scarring), limits the need for time off work and reduces overall costs.

This new ultrasound-guided surgical technique was tested on a series of 18 cadavers and then on a series of 15 patients for whom a lacertus syndrome had been diagnosed. The patients underwent the operation without any immediate surgical or anaesthetic complications. Muscle strength returned immediately and persisted. Pain was reduced and all patients who were working were able to carry out their professional activities from the very first week. The millimetric skin incision healed without hypertrophic scar tissue. A small haematoma appeared at week 1 and resolved spontaneously. No other late complications were observed.

In this context, this study would consolidate the preliminary results observed and confirm the hypothesis that minimally invasive percutaneous surgery under ultrasound is appropriate for sectioning Lacertus fibrosus safely, rapidly and effectively in Lacertus syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years and < 70 years
* Patient with isolated or bilateral Lacertus syndrome (no associated procedure on the day of surgery).
* Patient with a normal EMG

Exclusion Criteria:

* Patient with previous elbow surgery
* Patient with a history of elbow fracture
* Patient taking part in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disability and symptoms related to damage of the upper limb | Day 30
  Disability and symptoms will be assessed with Quick DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire (0 - 100 points). 0 means normal limb whereas 100 means full disability.

SECONDARY OUTCOMES:
Clamping force | Day 30 and Month 6
  Clamping force will be assessed with "key pinch " test. The pinch meter is placed between the tip of the thumb and the tip of the index finger. Result will be expressed in kilograms. Higher is weight, better is force.
Clamping force | Day 30 and month 6
  Clamping force will be assessed with Jamar test (grip test using a Jamar® hydraulic hand dynamometer). Result will be expressed in kilograms.Higher is weight, better is force.
Upper limb pain | Day1, Day 30 and month 6
  Upper limb pain will be assessed with VAS (Visual Analogic Scale) (0 - 10). 0 means no pain.
Persistent numbness | Day1, Day 30 and month 6
  Numbness will be assessed with VAS (Visual Analogic Scale) (0 - 10). 0 means no numbness whereas 10 means permanent numbness.
Patient satisfaction | Day 30 and month 6
  Satisfaction will be assessed with VAS (Visual Analogic Scale) (0 - 10). 0 means totally unsatisfied whereas 10 means totally satisfied.
Return to work | Day 30 and month 6
  Return to work will be assessed with "Return to work" date
Return to sport/artistic activities | Day 30 and month 6
  Return to sport/artistic activities with "Return to sport/artistic activities" date

CONTACTS AND LOCATIONS:
Overall Officials: Thomas APARD, MD, Principal Investigator — Clinique Les Franciscaines
Locations (1):
- Clinique Les Franciscaines, Versailles, Yvelines, France

IPD SHARING:
Plan to Share IPD: No